CLINICAL TRIAL: NCT06656676
Title: WePrEP: A Bilingual Shared Decision-making Tool to Facilitate Conversations Between Transgender Women and Their Providers as They Select an Ideal PrEP Method
Brief Title: WePrEP: Developing a PrEP Shared Decision-making Tool for Transgender Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Mile High Behavioral Healthcare Transgender Center of the Rockies (Unknown); The Gay Lesbian Bisexual & Transgender Community Center of Colorado (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH136932 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-10-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: HIV Prevention
Keywords: PrEP; Biomedical HIV prevention; CAB-LA; Cabenuva; Truvada; Tenofovir; oral PrEP; injectable PrEP; shared decision-making; transgender women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group: Transgender women (Experimental): Transgender women randomized to the intervention group will use WePrEP with a PrEP service provider. WePrEP will be stored on providers' tablets and will present oral PrEP and CAB-LA priority information points, identified during preliminary studies, and cue relevant discussions. Once a transgender woman assigned to the control group selects her preferred PrEP method, the provider will review the appropriate adherence strategies using WePrEP.
  Interventions: Behavioral: WePrEP: A shared decision-making tool
- Control group: Transgender women (Active Comparator): Transgender women randomized to the Control Group will receive a standard of care PrEP explanation from a PrEP services provider designated to deliver this trial condition. This explanation follows the 2021 CDC PrEP Clinical Guidelines, which have been updated to include information about CAB-LA.
  Interventions: Behavioral: Active comparator: CDC recommendations for discussing PrEP
- Intervention group: PrEP service providers (Experimental): During the study, PrEP service providers randomized to the intervention group will use WePrEP with transgender women participants in the intervention group who are potential PrEP patients. WePrEP will be stored on providers' tablets and will present oral PrEP and CAB-LA priority information points, identified during preliminary studies, and cue relevant discussions. Once the participant selects her PrEP method, the provider will review the appropriate adherence strategies. To ensure that they are able to provide feedback on WePrEP in IDIs, intervention group PrEP service providers will use WePrEP with a minimum of 8 different transgender women in this study.
  Interventions: Behavioral: WePrEP: A shared decision-making tool
- Control group: PrEP service providers (Active Comparator): PrEP service providers randomized to the Control Group will give transgender women enrolled in this study a standard of care PrEP explanation. This explanation follows the 2021 CDC PrEP Clinical Guidelines, which have been updated to include information about CAB-LA.
  Interventions: Behavioral: Active comparator: CDC recommendations for discussing PrEP

INTERVENTIONS:
Behavioral: WePrEP: A shared decision-making tool — WePrEP will be bilingual, both patient- and provider-facing, stored on the provider's electronic device (and will have the capability to integrate with electronic health records in the future to enable scalability), and easily accessible during in-person or virtual patient-provider encounters. WePrEP is designed to present pertinent PrEP information to transgender women and their PrEP service providers to stimulate discussions about PrEP choice and support adherence (once a PrEP strategy has been chosen). We hypothesize that this will ensure selection of the ideal PrEP method and improve subsequent adherence.
  Arms: Intervention group: PrEP service providers; Intervention group: Transgender women
Behavioral: Active comparator: CDC recommendations for discussing PrEP — Standard of care recommendations to discuss PrEP with potential end-users, endorsed by the CDC.
  Arms: Control group: PrEP service providers; Control group: Transgender women

SUMMARY:
HIV prevalence among transgender women (TW) in the United States is high (~14%). The best way to reduce HIV incidence in this population is to link TW to HIV pre-exposure prophylaxis (PrEP), which can reduce HIV transmission by up to 86%, with optimal adherence. The FDA approved the first long-acting form of PrEP, injectable cabotegravir (CAB-LA), in late 2021, which has the potential to decrease HIV transmission and increase PrEP adherence among TW. The addition of CAB-LA to available PrEP options necessitates TW and PrEP service providers select the best method (oral vs injectable) for each TW. However, TW have unique concerns about PrEP (e.g., interactions with gender-affirming hormones) and report that patient/provider discussions on this medication are suboptimal. Thus, to inform this shared decision process, the proposed study builds on formative work by developing and pilot-testing "WePrEP," a PrEP-focused bilingual digital shared decision-making tool (SDMT), tailored to diverse English- and Spanish-speaking TW and PrEP service providers. WePrEP will support communication between TW and PrEP service providers as they identify the ideal PrEP product for each TW and discuss associated adherence strategies by cuing conversations on TW's unique PrEP needs/concerns and presenting pertinent information that is culturally relevant and tailored to this population. To develop and test WePrEP, the investigators will partner with the Mile High Behavioral Healthcare Transgender Center of the Rockies, a Denver-based transgender-serving organization. They will use McNulty et al.'s adapted Shared Decision-Making Model for TW to guide the iterative participatory design process we will use with a group of racially/ethnically diverse TW and PrEP service providers, to develop WePrEP; we will begin this process using prototypes created from preliminary data (Aim 1a). The investigators will rigorously assess the usability of WePrEP via simulated patient/provider discussions (Aim 1b). Next, they will pilot test WePrEP in a randomized controlled trial (RCT; N=69 TW) with 2:1 randomization. In the RCT, PrEP service providers (N=4, of which n=1 is bilingual) will use WePrEP with intervention TW to select CAB-LA or oral PrEP and discuss adherence. Other providers (N=2, of which n=1 is bilingual) will give control TW a standard of care explanation of PrEP (CDC recommendations) to help them make their PrEP choice. TW will be referred to Sheridan Health Services to start PrEP. We will assess primary (feasibility; acceptability) and secondary (potential mechanisms of action of WePrEP; preliminary impact) outcome measures using validated scales and rigorous qualitative methods (Aims 2, 3). By creating a bilingual digital SDMT to enhance communication between TW and PrEP service providers as TW choose their ideal PrEP modality, this project is likely to make a widespread and lasting impact on TW's uptake and adherence to PrEP.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants in the transgender women group (N=69) must:

* Self-identify as a transgender woman (e.g., was assigned male at birth, but currently reports a feminine gender identity)
* Be between the ages of 18 and 65
* Currently live in the Denver area
* Speak English or Spanish
* Be HIV-negative (via Alere Determine)
* Not have participated in the development of WePrEP
* Not currently take PrEP, but report they are "interested in doing more to protect themselves from HIV" **We note that 1/3 of our RCT participants in the transgender women's group will be Black and/or Hispanic/Latina

Eligible participants in the PrEP service providers group (N=6) must:

* Not have participated in the development of WePrEP
* Live in the Denver area and (as a part of their employment responsibilities) discuss PrEP use with potential end-users.
* Have helped at least 1 TW make a decision about PrEP (e.g., whether or not to use it, which specific PrEP modality, etc...) in the last month.

Exclusion Criteria:

Participants in the transgender women group are excluded if they:

* Currently live with HIV
* Do not meet one or more of the inclusion criteria above

Participants in the PrEP service providers group are excluded if they:

* Do not live in the Denver area
* Do not meet one or more of the inclusion criteria above

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender women: defined as people assigned male at birth, but have a current feminine gender identity
Enrollment: 75 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility | At enrollment
  Feasibility of Intervention Measure (FIM) [Range: 1-5; Higher scores mean greater feasibility]
Acceptability | At enrollment
  Acceptability of Intervention Measure (AIM) [Range: 1-5; Higher scores mean greater acceptability]

SECONDARY OUTCOMES:
Preliminary impact (1st of 3 measures) | The proportion of transgender women who receive either form of PrEP is measured at enrollment.
  Proportion of transgender women who receive their first dose of either form of PrEP (measured at enrollment).
Preliminary impact (2nd of 3 measures) | For oral PrEP: PrEP serum concentrations are measured at 3 months. For injectable PrEP: PrEP serum concentrations are measured at 2 months.
  Proportion of transgender women who have a high enough serum concentration of either form of PrEP to prevent HIV at the second dose (measured at follow-up).
Preliminary impact (3rd of 3 measures) | For oral PrEP: PrEP refills are measured at 3 months. For injectable PrEP: Injections are measured at 2 months.
  Proportion of transgender women who refill (oral PrEP) or take an injection (injectable PrEP) at the second dose (measured at follow-up).
Mechanisms of action: Patient/provider communication (1st of 7 measures) | Measured at enrollment
  Communication composite measure from the Consumer Assessment of Healthcare Providers & Systems (CAHPS) [Range: 1-4; Higher scores mean better communication]
Mechanisms of action: Satisfaction with communication (2nd of 7 measures) | Measured at enrollment
  Combined Outcome Measure for Risk Communication and Treatment Decision-making Effectiveness (COMRADE) [Range: 1-5 where higher scores mean greater satisfaction]
Mechanisms of action: Patient/provider engagement (3rd of 7 measures) | Measured at enrollment
  Engagement with Health Care Providers (HCP) scale [Range: 1-5, where higher scores mean greater engagement]
Mechanisms of action: Evidence of shared decision-making (4th of 7 measures) | Measured at enrollment
  Control Preferences Scale (CPS) - domain measuring actual control over decision [Range: 1-5, where higher scores mean greater control]
Mechanisms of action: Satisfaction with control over PrEP decision (5th of 7 measures) | Measured at enrollment
  Control Preference Scale (CPS) - domain measuring control satisfaction [Range: 1-5, where higher scores mean greater satisfaction]
Mechanisms of action: Knowledge, motivation and self-efficacy to use PrEP (6th of 7 measures) | Measured at enrollment
  PrEP Knowledge, Motivation, & Self-Efficacy Assessment [Range: 1-5, where higher scores mean greater knowledge, motivation, and self-efficacy]
Mechanisms of action: Satisfaction with PrEP choice (7th of 7 measures) | Measured at follow-up (for oral PrEP users, this is at 3 months; for injectable PrEP users, this is at 2 months)
  Treatment Satisfaction Questionnaire [Range: 1-5, where higher scores mean greater satisfaction]

CONTACTS AND LOCATIONS:
Locations (1):
- Transgender Center of the Rockies, Sheridan, Colorado, United States

IPD SHARING:
Plan to Share IPD: No